CLINICAL TRIAL: NCT01713673
Title: Feasibility Study: A Prospective, Parallel, Randomized, Sham-controlled, Blinded Pilot Trial of the Safety and Efficacy of the Ulthera® System for Treatment of Axillary Hyperhidrosis
Brief Title: Feasibility Study: Safety and Efficacy of the Ulthera® System for Treatment of Axillary Hyperhidrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ULT-125
Record Dates: First submitted 2012-10-22; First posted 2012-10-25 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2013-06

CONDITIONS: Hyperhidrosis
Keywords: Hyperhidrosis; Axillary sweating; Ulthera® System; Ultherapy™ Treatment; Ulthera, Inc.
MeSH Terms: conditions — Hyperhidrosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Treatment (Experimental): Subjects receive Ulthera System Treatments according to the pre-defined Ulthera® System energy settings.
  Interventions: Drug: Ulthera System Treatment
- Sham Treatment (Sham Comparator): Subjects will receive Sham treatments using the Ulthera® System with the energy set to 0.00 Joules.
  Interventions: Drug: Sham treatment

INTERVENTIONS:
Drug: Ulthera System Treatment — Focused ultrasound energy delivered below the surface of the skin
  Other Names: Ultherapy™
  Arms: Active Treatment
Drug: Sham treatment — Study treatment using the Ulthera System, but delivering no ultrasound energy.
  Arms: Sham Treatment

SUMMARY:
Up to 20 subjects will be treated. Subjects will receive two (2) bilateral Ultherapy™ or Sham treatments of the axilla. The study hypothesis is that subjects who receive Ultherapy™ treatment will have a greater reduction in axillary sweating compared to subjects receiving Sham treatments. Follow-up visits will occur at 7 and 14 days following treatment #1, and at 7, 14, 30, 60 and 90 days following treatment #2. At each follow-up visit, assessments will be completed to compare the amount of axillary sweating compared to baseline.

DETAILED DESCRIPTION:
This study is a prospective, single-center, randomized, sham-controlled, blinded pilot clinical trial. Subjects will be randomly assigned to one of two treatment groups in a 2:1 randomization scheme, two (2) subjects assigned to receive Ultherapy™ treatment to every one subject assigned to receive Sham treatment.

Gravimetric measurement of sweat production and starch iodine tests will be performed, and Hyperhidrosis Disease Severity Scale (HDSS) scores will be obtained, prior to treatment and at each follow-up visit. Patient satisfaction will also be assessed. Sham treated subjects will have the option of continuing to Stage II and receive active treatment after completion of their Stage I 90 day study visit.

In a protocol amendment, the initial Stage I study cohort, excluding Sham treated subjects who opt to continue to Stage II, will be recruited to complete one long-term follow-up visit at 365 days following subjects' second study treatment. The same follow-up assessments will be completed to compare the amount of axillary sweating compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, ages 18-75
* Subject is in good health
* Diagnosis of bilateral axillary hyperhidrosis refractory to previous topical therapies
* At least 50 mg of spontaneous resting axillary sweat production in each axilla measured gravimetrically at room temperature/humidity over a period of 5 minutes
* A HDSS score is 3 or 4. An attempt will be made to approximate an equal number of scores 3 and 4
* Understands and accepts the obligation not to undergo any other procedures in the areas to be treated through the follow-up period
* Absence of physical conditions unacceptable to the investigator
* Willingness and ability to provide written informed consent and HIPAA authorization prior to performance of any study-related procedure
* Subjects of childbearing potential must have a negative urine pregnancy test result and must not be lactating

Exclusion Criteria:

* Dermal disorder including infection at anticipated treatment sites in either axilla
* Previous botulinum toxin treatment of the axilla in the past year
* Expected use of botulinum toxin for the treatment of any other disease during the study period
* Known allergy to starch powder or iodine
* Secondary hyperhidrosis, for example, hyperhidrosis that is secondary to other underlying diseases including hyperthyroidism, lymphoma and malaria
* Previous surgical treatment of hyperhidrosis including sympathectomy, surgical debulking of the sweat glands, subcutaneous tissue curettage and ultrasonic surgery
* Unwillingness to wash off deodorants and abstain use 72 hours prior to treatments or assessments
* History of previous Ultherapy™ treatment to the axilla
* Subjects with a history of a bleeding disorder
* Use of cholinomimetics, anticholinergics, or any oral herbal medicine treatments for hyperhidrosis
* Inability to withhold use of antiperspirants and deodorants, or any other topical treatments for hyperhidrosis within 72 hours prior to study treatments and assessments
* Unwillingness for complete shaving or removal of underarm hair within 12 hours prior to study treatments and follow-up visits

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-12; Primary Completion 2012-06 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with HDSS scores of 1 or 2 | 30 days post-treatment #2
  The HDSS scale is a qualitative measure of the severity of the condition based on how it affects subjects' daily activities. Subjects select the statement that best reflects their experience with underarm sweating on a 4 point scale, with 1 = sweating never noticeable and 4 = sweating is intolerable.

SECONDARY OUTCOMES:
Reduction in spontaneous axillary sweat production | Participants will be followed to 365 days post treatment #2
  Assessed by a gravimetric method as measured by a 50% reduction or more compared to baseline.
Subject Satisfaction | Participants will be followed to 365 days post-treatment #2
  Subject satisfaction will be measured using a Patient Satisfaction Questionnaire (PSQ.)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Nestor, MD, PhD, Principal Investigator — The Center for Clinical and Cosmetic Research
Locations (1):
- The Center for Clinical and Cosmetic Research, Aventura, Florida, United States